CLINICAL TRIAL: NCT05778240
Title: Behavioral Interventions to Increase Adherence to Palivizumab Prophylaxis in Children With Congenital Heart Disease: A Randomized Controlled Trial
Brief Title: Adherence to Palivizumab Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kosuyolu Heart Hospital (Other)
Collaborators: Sabanci University (Other); Maras Necip Fazil City Hospital (Unknown); Kocaeli University (Other); Van Research and Education Hospital (Unknown); Sakarya University (Other); Sivas Numune Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Erolu, Associate Professor, Kosuyolu Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020/14/413
Record Dates: First submitted 2023-02-17; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Congenital Heart Disease in Children; RSV

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Status quo bias and implementation intention bias (Experimental): Participants' families in this arm were informed about prophylaxis program and provided a schedule additionally called two days before appointments (status quo bias) and were asked to plan the appointment day (implementation intention).
  Interventions: Behavioral: Phone call
- Availability bias and social norm (Experimental): Participants' families in this arm were informed about prophylaxis program and provided a schedule and were received messages biweekly informing about benefits of program and adherence rate (availability bias and social norm).
  Interventions: Behavioral: Text message
- Control (Experimental): Participants' families in this arm were informed about prophylaxis program and provided a schedule
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Phone call — Participants were given the vaccination appointment card and participants received a telephone call every month two days before their appointment. Participants were reminded that they have a set appointment and were asked to plan the day of their appointment as detailed below. The standard script used in the telephone call in every hospital was as follows:Hello, we are calling you because you are enrolled in the palivizumab prophylaxis research program. As you know, you have a vaccination appointment on [enter date] at [enter time]. To help you plan your day of appointment, we have a few short questions.
  1. At your appointment day, will you be coming to the hospital from home, or will you need to get permission from your workplace?
  2. What kind of transportation do you plan to take to come to the hospital at your appointment day?
  3. At what time do you plan to leave home or work to come to the hospital?
  Arms: Status quo bias and implementation intention bias
Behavioral: Text message — Participants were given the vaccination appointment card and participants were included in a messaging group (on Whatsapp or SMS, depending on the participant's preference) where, twice a month they received a message informing them on RSV, on the additional risks caused by RSV infection in children with congenital heart diseases and on the benefits of adherence to the prophylaxis program. These messages also involved statements about the high number of patient families that kept their appointments in the previous month.
  Arms: Availability bias and social norm
Behavioral: Control — Participants were given the vaccination appointment card.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to analyze implications of two alternative nudge-interventions to increase adherence to palivizumab prophylaxis in children with congenital heart disease. The main questions investigators aim to answer are:

* Are well-established cognitive biases effective in increasing patient families' adherence to the palivizumab prophylaxis program?
* What are the factors that affect families' adherence to the prophylaxis program and whether and how the effects of interventions depend on these factors?

To study these questions investigators planned to utilize four well-established cognitive biases in designing two alternative nudge-interventions and investigators measured the effectiveness of each nudge-intervention against a control group.

Patients were randomly allocated to one control and two treatment groups. In the control group, investigators informed participants about the prophylaxis program and provided a schedule. Patients in the first treatment group were additionally called two days before appointments (status quo bias), and were asked to plan the appointment day (implementation intention). Patients in the second treatment group received biweekly messages informing them about the benefits of the program as well as the current adherence rate (availability bias and social norm).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital heart disease which are hemodynamically unstable, congestive heart failure, diagnosis of congenital heart disease with hemodynamically significant residual defects after corrective heart surgery, cardiomyopathy, pulmonary hypertension
* Being between 0-2 years of age

Exclusion Criteria:

* Diagnosis of congenital heart disease in which palivizumab prophylaxis is not needed (the diagnosis of congenital heart diseases which are hemodinamically stable.)
* Becoming exitus during prophylaxis program
* Not being between 0-2 years of age

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 229 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of cognitive biases in increasing adherence to prophylaxis programme | 4 weeks
  The average adherence rates in the control and treatment groups

SECONDARY OUTCOMES:
The effect of father employment status (full-time, part-time, no) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of number of children in the family on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of birth weight (weight in grams) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of number of intensive care unit admissions on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of knowledge about respiratory syncytial virus previously (yes/no) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of finding prophylaxis program important or not (yes/no) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of the distance between home and hospital (km) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of number of difficulties about accessing to prophylaxis program on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of family size (number of people living in the same house) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of the number of children in the school age on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of family income (<1000 TL, 1000-2999 TL, 3000-4999 TL, 5000-6999 TL, 7000-8999 TL, >9000 TL ) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of smoking (yes/no) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of father and mother's age (years) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of father and mother education level (no education, primary school, high school, university) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of employment status of mother on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of marital status (married, married- separated, divorced, widowed) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.
The effect of health status of father and mother (in good health, in moderate health, in bad health) on the participants' adherence to the prophylaxis program | 8 weeks
  Factor that affects participants' adherence to the prophylaxis program. The interaction of each factor on the treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Erolu, M.D.Ph.D., Principal Investigator — Kosuyolu Heart Hospital
Locations (1):
- Kosuyolu Heart Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erolu E, Kibris O, Tosun Y, Yildirim A, Pamukcu O, Basar EZ, Babaoglu K, Epcacan S, Donmez Y, Giray D, Dervisoglu P, Tasci O. Behavioural interventions to increase adherence to palivizumab prophylaxis in children with CHD. Cardiol Young. 2024 Apr 26:1-8. doi: 10.1017/S1047951124024946. Online ahead of print. PMID 38664919